CLINICAL TRIAL: NCT04792034
Title: An Open-label, Two-Arm, Pharmacokinetics, Safety, and Tolerability Study of a Single Topical Dose of GOPRELTO® Nasal Solution and a Single Dose of NUMBRINO™ Nasal Solution for the Induction of Local Anesthesia of the Mucous Membranes When Performing Diagnostic Procedures and Surgeries in Pediatric Subjects From ≥12 Years to <18 Years of Age
Brief Title: Pharmacokinetics, Safety, and Tolerability Study of GOPRELTO® Nasal Solution and NUMBRINO™ Nasal Solution
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Noden Pharma (Industry)
Collaborators: Omnivium Pharmaceuticals LLC (Industry); LXO Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RA-VP-000-357; NCT07287735 (obsolete NCT alias)
Record Dates: First submitted 2021-02-22; First posted 2021-03-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: ENT Disorder; Nasal Procedures; Nasal Anesthesia; Nasal Mucosa Surgery
Keywords: Nasal; Sinus; ENT
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Intervention Model Description: Open-label, single-dose, non-randomized, two-arm sequential, single-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GOPRELTO® nasal solution, 4%, (Experimental): FDA Approved GOPRELTO® (cocaine hydrochloride nasal solution, 4%); Up to 160 mg depending on subject's weight; Saturated cottonoid pledgets are applied topically in both nostrils by study personnel
  Interventions: Drug: Cocaine Hydrochloride Nasal Solution
- NUMBRINO™ nasal solution, 4% (Experimental): FDA Approved NUMBRINO™ (cocaine hydrochloride nasal solution, 4%); Up to 160 mg depending on subject's weight; Saturated cottonoid pledgets are applied topically in both nostrils by study personnel
  Interventions: Drug: Cocaine Hydrochloride Nasal Solution

INTERVENTIONS:
Drug: Cocaine Hydrochloride Nasal Solution — Topical Anesthetic
  Other Names: GOPRELTO®
  Arms: GOPRELTO® nasal solution, 4%,
Drug: Cocaine Hydrochloride Nasal Solution — Topical Anesthetic
  Other Names: NUMBRINO™
  Arms: NUMBRINO™ nasal solution, 4%

SUMMARY:
The purpose of this study is to assess the pharmacokinetic (PK) properties, safety and tolerability following a single dose administration of GOPRELTO® or NUMBRINO™ as an anesthetic for diagnostic procedures and surgeries on or through the mucous membranes of the nasal cavities in pediatric adolescent subjects.

DETAILED DESCRIPTION:
GOPRELTO® and NUMBRINO™ (cocaine hydrochloride nasal solution, 4%) are approved anesthetic products in adults. The purpose of this study is to assess the pharmacokinetic (PK) properties, safety, tolerability, and dosing of GOPRELTO® and NUMBRINO™ each as an anesthetic for diagnostic procedures and surgeries on or through the mucous membranes of the nasal cavities in pediatric adolescent subjects.

The primary objectives for each treatment of the study are:

* To assess the safety and tolerability of GOPRELTO® and NUMBRINO™ nasal solution in pediatric adolescent subjects as an anesthetic for diagnostic procedures and surgeries on or through the mucous membranes of the nasal cavities, respectively.
* To evaluate the PK properties and define the dosing for GOPRELTO® and NUMBRINO™ nasal solution, respectively, in pediatric adolescent subjects as an anesthetic for diagnostic procedures and surgeries on or through the mucous membranes of the nasal cavities.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in the study if he or she meets all of the following criteria:

1. Is accompanied and/or represented by a parent or guardian able to comprehend and sign the informed consent document.
2. Is able to understand and provide assent to an age-appropriate subject assent form (as defined by local practice or regulation).
3. Subject or parent/guardian is able to communicate with the Investigator and comply with the requirements of the protocol.
4. Is male or female ≥12 to <18 years of age at the time of dosing.
5. Is no lower than the 10th percentile for weight according to age.
6. Has a body mass index (BMI) no lower than the 5th percentile by age.
7. Has an oxygen saturation of at least 98%.
8. Will be undergoing a diagnostic procedure or surgery on or through the nasal mucous membranes of either one or both nostrils.
9. Is a non-pregnant, non-lactating female (if of child-bearing potential and sexually active) or is a male (if sexually active with a partner of child-bearing potential) who agrees to use a medically acceptable and effective birth control method from the time of the Screening Visit and then for 8 days following the last dose of GOPRELTO® nasal solution or NUMBRINO™ nasal solution administration. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include: abstinence, FDA-approved hormonal contraceptives (i.e., birth control pill, injection, patch or vaginal ring), diaphragm, intrauterine device, double-barrier methods, surgical sterilization, and progestin implant or injection. Prohibited methods include: the rhythm method or withdrawal.

Exclusion Criteria:

A subject will be excluded from the study if he or she meets any of the following criteria:

1. Has a history of seizure.
2. Has a known hypersensitivity allergy to any ester-based anesthetics including cocaine hydrochloride, procaine, tetracaine, chloroprocaine, dibucaine, or benzocaine, and/or any other compounds of the drugs and /or devices that are part of this protocol (amide based anesthetics are NOT exclusionary).
3. Has previously received intranasal topical cocaine within 14 days prior to the Screening Visit.
4. Has participated in an investigational study or received an investigational drug within 30 days preceding Treatment Day 1.
5. Has a history of abuse of controlled substances, nasal or otherwise.
6. Has a positive test result for drugs of abuse at the Screening Visit: amphetamines, barbiturates, cannabinoids, cocaine metabolites, opiates, and oxycodone via a urine test. Alcohol is prohibited within 24 hours prior to Treatment Day 1.
7. Is a pregnant female or nursing mother or has a positive urine pregnancy test at the Screening Visit or on Treatment Day 1.
8. Use of any serotonin-norepinephrine reuptake inhibitors/selective serotonin reuptake inhibitors (SNRIs/SSRIs) up to 14 days prior to the Screening Visit or has a need to use these drugs at any time throughout the duration of the study.
9. Use of monoamine oxidase inhibitor (MAO) drugs up to 14 days prior to the Screening Visit or has a need to use these drugs at any time throughout the duration of the study.
10. Use of nasal products such as decongestants (oxymetazoline, phenylephrine), amphetamines, stimulant prescription and nonprescription products such as catecholamines (direct and indirect-acting sympathomimetics), bronchial inhalers containing sympathomimetics (epinephrine or other beta-receptor agonists), or herbal products in the 2 days prior to the Screening Visit or has a need to use these drugs through or on Treatment Day 1.
11. Use of disulfiram.
12. Planned or anticipated need for additional vasoconstrictor agents such as epinephrine or phenylephrine.
13. Suffers from a condition, other than the need for a diagnostic procedure or surgery on or through the nasal mucous membranes, which in the opinion of the Investigator, would compromise the safety of the subject, the quality of the data, or the normal wound healing process.
14. Has severely traumatized mucosa or septum in the nasal cavities or has damage to the nasal space that will not allow pledgets to be inserted.
15. Has a recent or active history of myocardial infarction, coronary artery disease, congestive heart failure, unstable angina, or uncontrolled hypertension. Uncontrolled hypertension is defined as systolic blood pressure or diastolic blood pressure greater than or equal to the 95th percentile by sex, age and height.
16. Has an ECG finding of any abnormality at the Screening Visit. Generally, these exclusionary abnormalities are current or prior myocardial ischemia or infarction, dysrhythmia, or risk of serious dysrhythmia (such as prolonged QT interval). An exception to this would be if sinus bradycardia or sinus tachycardia is present. The Investigator must determine whether this finding is clinically significant and exclusionary.
17. Has a known personal or family history of hereditary pseudocholinesterase deficiency.
18. Has a known or suspected personal or family history of pheochromocytoma. Study participants will be specifically asked if they have been treated for a pheochromocytoma previously or if they have a family member who has been diagnosed with pheochromocytoma (as 10% of these are familial).
19. Has any laboratory result outside the normal laboratory reference range deemed clinically significant by the Investigator.
20. Has a history of, or current, hepatic or renal disease.
21. Is not suitable for entry into the study, in the opinion of the Investigator. Note: A one-time retest is permitted for any blood test if the original sample was hemolyzed.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Blood pressure | Baseline and every 5 minutes through 90 minutes post-pledget application.
  Changes in blood pressure from baseline of 20 mmHg systolic or 15 mmHg diastolic OR when blood pressure reaches 150/90 mmHg in the automated blood pressure monitoring system during the mentioned time frame.
  Measurements will be taken in supine position with 3 measurements 5-6 minutes apart.
Changes in Heart rate | Baseline and every 5 minutes through 90 minutes post-pledget application.
  Increase in heart rate from baseline of 20 bpm OR when heart rate of 125 bpm is reached at any point in the automated vital sign monitoring system during the mentioned time frame.
Changes in Respiratory Rate | Baseline and every 15 minutes through 90 minutes post-pledget application.
  Any changes in respiratory rate (increase or decrease) while on study medication.
Physical examination | Screening Visit
  Assessment of skin, head, ears, eyes, nose, throat, neck, thyroid, lungs, heart, cardiovascular, abdomen, lymph nodes, and musculoskeletal system/extremities; oral temperature, height, weight; BMI as well as height and weight percentiles.
Electrocardiogram | Screening Visit, and on Day 1 at Baseline (pre-dose), continuously during treatment, and through 90 minutes post-pledget application
  Any changes or delays in heart rhythm while on medication. Electrocardiogram will be performed in the supine position.
Pulse Oximetry | Screening Visit, and on Day 1 at Baseline (pre-dose), continuously during treatment, and through 90 minutes post-pledget application
  Any changes in the amount of oxygen in the blood while on study medication.
Incidence of Adverse events (AEs) | From Day 1 (pledget application) through the final follow-up call at Day 10.
  The number and percentage of subjects with AEs, AEs severity, causality, Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs).
Maximum observed plasma concentration (Cmax) | Screening Visit, Baseline (pre-dose), 20, 40, 60, and 90 minutes, and 2, 4, and 8 hours after pledget application.
  Measurement of the amount of the study medication (cocaine topical solution) in the blood over 8 hours to define the Cmax.
Time to maximum observed plasma concentration (Tmax) | Screening Visit, Baseline (pre-dose), 20, 40, 60, and 90 minutes, and 2, 4, and 8 hours after pledget application.
  Measurement of the time it takes after dosing for the study medication (cocaine topical solution) to reach its highest observed concentration in the blood over 8 hours.
Area under the plasma concentration versus time curve from time of dosing (0) to the time of last quantifiable concentration (AUClast) | Screening Visit, Baseline (pre-dose), 20, 40, 60, and 90 minutes, and 2, 4, and 8 hours after pledget application.
  Measurement of the amount of the study medication (cocaine topical solution) in the blood over 8 hours to define the AUC.
Area under the plasma concentration versus time curve from time of dosing (0) to infinity (AUCinf) | Screening Visit, Baseline (pre-dose), 20, 40, 60, and 90 minutes, and 2, 4, and 8 hours after pledget application.
  Measurement of the total exposure to the study medication in the blood over 8 hours, starting from dosing and extrapolated to infinity.
Terminal rate constant in plasma from the negative of the regression line slope through the ln plasma concentration versus time data defining the terminal phase [kel (λz)] | Screening Visit, Baseline (pre-dose), 20, 40, 60, and 90 minutes, and 2, 4, and 8 hours after pledget application.
  Measurement of the time it takes for the concentration of the study medication in the blood to decrease by half during the terminal elimination phase, over 8 hours, calculated using kel as ln(2)/kel.
Terminal half-life in plasma calculated from the kel as ln(2)/kel (t½) | Baseline (pre-dose), 20, 40, 60, and 90 minutes, and 2, 4, and 8 hours after pledget application.
  Measurement of the rate at which the study medication is eliminated from the blood during the terminal phase, calculated from the slope of the log-transformed concentration versus time data.

OTHER OUTCOMES:
Application Site Assessment | Screening Visit, Day 1 before drug application (Baseline), and within 90 minutes following the completion of the procedure.
  A visual nasal examination to determine if irritation is present at the application site.
Pediatric Smell Wheel | Screening Visit and 90 minutes post-procedure on Day 1.
  Assessment of smell (pre-dose and post-dose smell tests).
Assessment of Analgesia and Anesthesia | Screening Visit and on Day 1 (following pledget removal but prior to procedure).
  Assessment of analgesia and anesthesia will be conducted using a monofilament (Von Frey filament).
Pledget size assessment | Screening Visit and Day 1 (pre-dose).
  A pledget size assessment will be conducted to assess the appropriate size pledget to administer study drug.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - SCENT Sleep and Allergy, 110 Highland Center Drive, Columbia, South Carolina
  - SCENT Sleep and Allergy, 145 Park Central, Columbia, South Carolina
  - South Carolina ENT, Sleep and Allergy, Columbia, South Carolina
  - SCENT Sleep and Allergy, 15 Exchange Dr., Lugoff, South Carolina

IPD SHARING:
Plan to Share IPD: No